CLINICAL TRIAL: NCT03799237
Title: Cluster Randomized Controlled Trial: Efficacy of Gravid Oviposition Sticky Trap (GOS) and Dengue NS1 Antigen Rapid Diagnostic Test for Early Surveillance of Dengue Among Adult Aedes Mosquitoes to Reduce Dengue Outbreaks in PJU10, Damansara Damai, Selangor, Malaysia
Brief Title: Combating Dengue With Innovative, Paradigm-shift-Strategies: Early Dengue Surveillance in Adult Aedes Mosquitoes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jonathan Liew Wee Kent (Other)
Collaborators: Petaling Jaya City Council, Malaysia (Unknown); Selangor State Health Department, Malaysia (Unknown)
Responsible Party: Sponsor-Investigator, Jonathan Liew Wee Kent, Postdoctoral Research Fellow, University of Malaya
Organization: University of Malaya (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GOSNS1-1; MO013-2017 (Other Grant/Funding Number: Malaysia Ministry of Education)
Record Dates: First submitted 2019-01-02; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Dengue
Keywords: Dengue; Adult Aedes; GOS trap; Dengue NS1 antigen test; Early dengue detection and surveillance
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GOS trap and dengue NS1 antigen kit (Experimental): Gravid Oviposition Sticky (GOS) traps will be placed to trap adult Aedes mosquitoes and changed weekly. NS1 will be used to detect dengue in trapped Aedes mosquitoes. When dengue NS1 positive mosquitoes are found, community will be alerted via flyers, banners and other means. Routine Aedes/dengue control and surveillance will be carried out as usual as per the current Ministry of Health guidelines.
  Interventions: Other: GOS trap and dengue NS1 antigen kit
- Control (No Intervention): The GOS traps will be placed randomly in the control arm once per month for entomological survey. Routine Aedes control and surveillance will be carried out as per the current Ministry of Health guidelines. Dengue control measure will be initiated by the health authorities when human cases are reported from this arm.

INTERVENTIONS:
Other: GOS trap and dengue NS1 antigen kit — The GOS trap lure and sticky surfaces to trap gravid Aedes mosquitoes. Three GOS traps will be placed on every 3 floors of the residential blocks. The traps will be changed weekly. Trapped Aedes mosquitoes will be identified to species. The mosquitoes will then be dissected, to remove the abdomen from the thorax. Five to seven abdomens of the same mosquito species will be pooled and tested for dengue NS1 antigen using the SD Biosensor Standard Q dengue NS1 antigen test kit. If the pool is tested positive for dengue NS1, the head and thorax of the respective abdomens will be subjected to the same procedure for dengue NS1 antigen test, individually. This may allow us to identify a focus where there could be dengue-infected individuals. Flyers/Posters will be disseminated besides, house-to-house approach to inform the residents of the findings and apartment blocks where these mosquitoes were found. The apartment management will also make use of social media disseminate this information.
  Arms: GOS trap and dengue NS1 antigen kit

SUMMARY:
During dengue outbreaks, the Ministry of Health Malaysia employs various methods to control the spread of disease, including killing the larvae of Aedes mosquitoes, fogging, together with educating and disseminating information about the dengue outbreak, to the community. However, this is too late. Research has shown that when an outbreak has occurred, the viral infection has already spread among the community. Therefore, this current trial aims to educate the public (via questionnaire survey and interactions with the residential managements, mainly), detect dengue-infected mosquitoes, inform the communities of the presence of dengue-infected mosquitoes, followed by approaching and educating them to take precautionary measures before the outbreak happens. Trapping (using gravid oviposition sticky (GOS) traps) and detecting dengue virus non-structural 1 (NS1) antigen (using dengue NS1 kit) in the Aedes mosquitoes will be a more reliable way to alert the community before a potential dengue outbreak in their housing area. The community will receive information of presence of infected mosquitoes and probable dengue infections before dengue cases are reported. This will be an ideal time for clean-ups and for search and destroy activities. With this shift in approach and the use of newer techniques, it is hoped that deaths and epidemics due to dengue will be reduced.

DETAILED DESCRIPTION:
This cluster randomised controlled trial will be conducted to provide evidence on the efficacy of an integrated active vector surveillance and preventive strategy in the community. It aims to demonstrate effectiveness of a new proactive paradigm in reducing dengue epidemics. The main hypotheses are 1) This new paradigm (GOS trap and dengue NS1 kit for detection of dengue in Aedes) will reduce dengue epidemics compared to the usual current vector surveillance/control carried out by the Ministry of Health. 2) Community will be more receptive to this new surveillance activity as they will receive information of dengue transmissions before dengue cases are reported.

The study sites at PJU10, Damansara Damai, Petaling Jaya, Selangor, Malaysia are

1. Intervention arm: Harmoni Apartment, Impian Apartment, Park Avenue Condominium, and Suria Shop Apartment
2. Control arm: Permai Apartment, Lestari Apartment, Indah Apartment, and Vista Shop Apartment

Activities to be carried out include:

A. Questionnaire survey and blood taking for dengue seroprevalence among residents from both arms When people in the community are gathered at an identified, suitable area, the Knowledge, Attitude and Practice (KAP) questionnaires will be distributed for them to answer. After the questionnaire survey, about 3 ml of venous blood would be taken by trained personnel for dengue IgG and IgM serology.

B. Placement of the GOS mosquito trap in the intervention arm The GOS mosquito traps will be placed in the intervention arm and serviced weekly. The trapped Aedes mosquitoes would be checked for dengue virus via dengue NS1 rapid diagnostic test kit.

The GOS mosquito traps will also be placed randomly in the control arm once per month for entomological survey.

C. If a dengue-positive mosquito is found, flyers and banners will be distributed and hung to inform the residents of the presence of dengue transmission in the apartment block/apartment. Alternatively, the residents may also be approached house-to-house or an educational booth set up at strategic locations in the apartment to warn and educate the residents.

D. The KAP questionnaire survey will be carried out again 3 months before the completion of the trial in the intervention arm to gauge the communities' perception of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above, including pregnant women and healthy individuals
* Reside in the study sites
* Work at the study sites for at least 40 hours per week
* Able to give consent
* Willing to participate in blood taking

Exclusion Criteria:

* Age below 18 years
* Unable to give consent
* Not willing to undergo venepuncture or finger-prick

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7979 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in number of weekly notified dengue cases in intervention arm | Assess weekly, through study completion, 1 and a half years
  The number of notified dengue cases in the study sites will be obtained from the District Health Office
Change in the duration of dengue outbreaks in intervention arm | Through study completion, an average of 1 and a half years
  The duration of dengue outbreaks in the study sites will be obtained from the District Health Office.

SECONDARY OUTCOMES:
Change in adult Aedes density in the intervention arm | Assess weekly, through study completion, within 1 and half years.
  Based on the weekly trap index
Change in level of dengue Knowledge, Attitude and Practice in the intervention arm | 6 months after recruitment for pre-trial questionnaire survey. 3 months after recruitment for post-trial questionnaire survey, through study completion, 1 and a half years
  The mean of the percentage score of the population for each domain (knowledge & attitude/practises) will be determined for the pre- and post-test. Then, paired t-test will be performed to determine the presence of significant changes in both means (An increase in score percentage indicate a better outcome). Additionally, an individual percentage score of 80% and above indicates indicates good knowledge/attitude/practice.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan WK Liew, PhD, Principal Investigator — University of Malaya; Indra Vythilingam, PhD, Study Director — University of Malaya
Locations (1):
- Petaling Jaya City Council, Petaling Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No
Medical ethics have been obtained with a statement that these information is confidential. These information will be deleted within 1 year after the study is completed

REFERENCES:
- [Background] Lau SM, Chua TH, Sulaiman WY, Joanne S, Lim YA, Sekaran SD, Chinna K, Venugopalan B, Vythilingam I. A new paradigm for Aedes spp. surveillance using gravid ovipositing sticky trap and NS1 antigen test kit. Parasit Vectors. 2017 Mar 21;10(1):151. doi: 10.1186/s13071-017-2091-y. PMID 28327173
- [Background] Klungthong C, Manasatienkij W, Phonpakobsin T, Chinnawirotpisan P, Rodpradit P, Hussem K, Thaisomboonsuk B, Ong-ajchaowlerd P, Nisalak A, Kalayanarooj S, Buddhari D, Gibbons RV, Jarman RG, Yoon IK, Fernandez S. Monitoring and improving the sensitivity of dengue nested RT-PCR used in longitudinal surveillance in Thailand. J Clin Virol. 2015 Feb;63:25-31. doi: 10.1016/j.jcv.2014.12.009. Epub 2014 Dec 12. PMID 25600599
- [Background] Roslan MA, Ngui R, Vythilingam I, Sulaiman WYW. Evaluation of sticky traps for adult Aedes mosquitoes in Malaysia: a potential monitoring and surveillance tool for the efficacy of control strategies. J Vector Ecol. 2017 Dec;42(2):298-307. doi: 10.1111/jvec.12270. PMID 29125255
- [Background] Chadee DD, Ritchie SA. Efficacy of sticky and standard ovitraps for Aedes aegypti in Trinidad, West Indies. J Vector Ecol. 2010 Dec;35(2):395-400. doi: 10.1111/j.1948-7134.2010.00098.x. PMID 21175947
- [Background] Gama RA, Silva EM, Silva IM, Resende MC, Eiras AE. Evaluation of the sticky MosquiTRAP for detecting Aedes (Stegomyia) aegypti (L.) (Diptera: Culicidae) during the dry season in Belo Horizonte, Minas Gerais, Brazil. Neotrop Entomol. 2007 Mar-Apr;36(2):294-302. doi: 10.1590/s1519-566x2007000200018. PMID 17607465
- [Background] Lee C, Vythilingam I, Chong CS, Abdul Razak MA, Tan CH, Liew C, Pok KY, Ng LC. Gravitraps for management of dengue clusters in Singapore. Am J Trop Med Hyg. 2013 May;88(5):888-892. doi: 10.4269/ajtmh.12-0329. Epub 2013 Mar 11. PMID 23478581
- [Background] Lau SM, Vythilingam I, Doss JI, Sekaran SD, Chua TH, Wan Sulaiman WY, Chinna K, Lim YA, Venugopalan B. Surveillance of adult Aedes mosquitoes in Selangor, Malaysia. Trop Med Int Health. 2015 Oct;20(10):1271-80. doi: 10.1111/tmi.12555. Epub 2015 Jul 14. PMID 26094839
- [Derived] Liew JWK, Selvarajoo S, Tan W, Ahmad Zaki R, Vythilingam I. Gravid oviposition sticky trap and dengue non-structural 1 antigen test for early surveillance of dengue in multi-storey dwellings: study protocol of a cluster randomized controlled trial. Infect Dis Poverty. 2019 Sep 3;8(1):71. doi: 10.1186/s40249-019-0584-y. PMID 31477185

DOCUMENTS (2):
  • Informed Consent Form (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT03799237/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-01-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT03799237/Prot_SAP_001.pdf